CLINICAL TRIAL: NCT00246272
Title: An Open-label Study Evaluating the Maintenance of Clinical Effect in Adults With Schizophrenia Switched From RISPERDAL® Tablets (Risperidone) to an Equivalent Dose of a Rapidly-dissolving Tablet Formulation of Risperdone
Brief Title: An Open-label Study Evaluating the Maintenance of Clinical Effect in Adult Schizophrenia Patients Switched From Risperidone Tablets to an Equivalent Dose of a Rapidly-dissolving Tablet Formulation of Risperdone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Ortho Inc., Canada (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR005956
Record Dates: First submitted 2005-10-28; First posted 2005-10-31 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2010-04

CONDITIONS: Schizophrenia
Keywords: risperidone; schizophrenia; rapidly-dissolving
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone

INTERVENTIONS:
Drug: risperidone

SUMMARY:
The purpose of this study is to evaluate the maintenance of clinical effect of a rapidly-dissolving tablet form of risperidone (an antipsychotic medication) in adult schizophrenia patients switched from their previous equivalent dose of RISPERDAL® tablets

DETAILED DESCRIPTION:
This trial is a non-randomized, open-label, single arm, multicentre study aimed at evaluating the maintenance of clinical effect of the rapidly-dissolving tablet dosage form of risperidone, in patients switched from their previous equivalent dose of conventional risperidone tablets (doses of 0.5 mg, 1 mg, 2 mg, 3 mg or 4 mg/day). Approximately 100 adult schizophrenia patients (ages >= 18 years) who are symptomatically stable will be enrolled. Patients will be asked to take an equivalent dose of the rapidly-dissolving tablet form of risperidone for 4 weeks of treatment. Other psychotropic medications taken at study entry may be continued throughout the study, providing the dose was stable prior to entry for a minimum of 4 weeks and will remain stable throughout the course of the study. Dose escalation/reduction of rapidly-dissolving risperidone tablets is not permitted. Study visits will take place twice over the 4 week period, once at study entry and again at the final visit. The primary efficacy parameter will be the CGI-Severity (CGI-S) score for maintenance of clinical effect. Secondarily, two 5-point Likert scales will be completed, one measuring clinician's assessment of anxiety symptoms and the other measuring clinician's assessment of depressive symptoms. Patients with existing symptoms of psychosis will be clinician rated on a 5-point Likert scale. Other secondary assessments include: Visual Analogue Scale (VAS) for risperidone acceptability, completed by the patient or the caregiver (if applicable). For each subject, the VAS score will be calculated on a 10 cm line ranging from a score of "0" (not acceptable) to "10" (very acceptable). Safety evaluations during the study will include vital signs and physical examination, body weight, adverse event surveillance, and urine pregnancy tests for females of childbearing potential. The study hypothesis is that the clinical effect will be maintained when schizophrenia patients previously stabilized on risperidone conventional tablets are treated with rapidly-dissolving risperidone tablets, and that risperidone rapidly dissolving tablets will be well tolerated.

Subjects who are stable on conventional risperidone tablets (0.5, 1, 2, 3 or 4 mg/day) for at least 2 weeks will be switched to an equivalent dose of rapidly-dissolving risperidone tablets (0.5, 1, 2, 3 or 4 mg/day). The study medication will be taken orally for 4 weeks, using the same frequency of dosing (once-daily, twice-daily, etc.) as with their previous conventional tablet regimen.

ELIGIBILITY:
Inclusion Criteria:

* Baseline CGI-Severity score of either "1" (not ill), "2" (very mildly ill), or "3" (mildly ill)
* Must have been on a stable dose of conventional risperdone tablets (doses of 0.5, 1, 2, 3 or 4 mg/day) to treat their disorder for a minimum of 2 weeks
* Patients must be able to comply with the study visit schedule and the patient (or a caregiver having frequent contact with the patient) must be able to complete the protocol specified assessments and trial questionnaires
* Females must be postmenopausal, surgically sterile, or practicing an effective method of birth control, and must have a negative urine pregnancy test pre-study and at the final visit
* Patient is otherwise healthy on the basis of a pre-trial physical examination and medical history

Exclusion Criteria:

* Patients who cannot take aspartame (an artificial sweetener that is a source of phenylalanine)
* Currently taking carbamazepine
* Have a history of neuroleptic malignant syndrome or other serious or unstable medical illnesses
* Females who is pregnant or breastfeeding
* Patients who have used an experimental drug or an experimental medical device within 30 days before the start of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2004-10; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
CGI-Severity (CGI-S) score for maintenance of clinical effect

SECONDARY OUTCOMES:
Separate 5-point Likert scales for clinician's assessment of (1) anxiety, (2) depressive, and (3) psychotic symptoms. Visual Analogue Scale (VAS) measurements for patient/caregiver acceptability of rapidly-dissolving risperidone will be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Ortho Inc. Clinical Trial, Study Director — Janssen-Ortho Inc., Canada